CLINICAL TRIAL: NCT02825407
Title: Creation et Characterization of Two Groups of Elderly Subjects so as to Evaluate the Link Between the Characteristics of Oral Physiology, Sensory Sensitivity, the Release in Vivo Aromatic Compounds, and In-mouth Comfort During the Consumption of Foods
Brief Title: Creation and Characterization of Two Groups of Subjects to Evaluate Sensitivity
Acronym: ALIMASSENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: VAN WYMELBEKE ANR 2014
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-06

CONDITIONS: Sensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Functional Status

ARMS (1):
- main study (Experimental)
  Interventions: Dietary Supplement: Oral physiology

INTERVENTIONS:
Dietary Supplement: Oral physiology

SUMMARY:
There are few data on elderly people concerning mechanisms involved in the in vivo release and perception of aromatic compounds. Any knowledge on this point would be of great interest to the scientific community. Concerning the dimensions of sensory perception and in-mouth comfort, there is, to our knowledge, no methodology to describe them. These dimensions are truly original and innovative, and investigating them will lead to the development of foods adapted to elderly populations with chewing and salivation disorders.

The expected results are:

* to obtain two groups of subjects with differences in chewing abilities and saliva production
* the characterization of flavour release profiles in elderly subjects with regard to oral physiology (mastication and salivation) and saliva composition
* a sensory profile describing in-mouth comfort when food is eaten

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written consent
* Age >= 65 years
* Persons living at home or in an old-people's home (Etablissement Hébergement Personnes Agées Dépendantes : EHPAD)
* Persons able to move around independently

Exclusion Criteria:

* Persons without national health insurance cover
* Persons in hospital
* Persons whose MMSE (Mini-Mental State Examination) is < 24
* Persons requiring enteral or parenteral feeding
* Persons who in the last 12 months have received € 4500 by participating in clinical studies, including the present study
* Persons in a period of exclusion following a previous study
* Food allergies
* Adults under guardianship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Dental health evaluation : GOHAI questionnaire (Geriatric Oral Health Assessment Index | At inclusion

SECONDARY OUTCOMES:
Measure of chewing efficacy : fast test of chewing, Masticatory Normality Index (MNI) | At inclusion

OTHER OUTCOMES:
Measure of salivary flows in the rest and in stimulation | Day 0 and month 9
Measure of strength of compression between the tongue and palate with the IOPI system | month 9
Volume of the oral cavity by acoustic reflectometry by means of a rhynopharyngometer | month 9

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Champmaillot Geriatric Department, Dijon, France